CLINICAL TRIAL: NCT02924727
Title: A Multi-center, Randomized, Double-blind, Active-controlled, Parallel-group Phase 3 Study to Evaluate the Efficacy and Safety of LCZ696 Compared to Ramipril on Morbidity and Mortality in High Risk Patients Following an Acute Myocardial Infarction (AMI)
Brief Title: Prospective ARNI vs ACE Inhibitor Trial to DetermIne Superiority in Reducing Heart Failure Events After MI
Acronym: PARADISE-MI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLCZ696G2301; 2016-002154-20 (EudraCT Number)
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Acute Myocardial Infarction
Keywords: Spontaneous AMI; HF hospitalization; outpatient HF; LV systolic dysfunction; pulmonary congestion; STEMI; NSTEMI; randomized clinical trial; LCZ696; ramipril
MeSH Terms: conditions — Ventricular Dysfunction, Left; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction | interventions — sacubitril and valsartan sodium hydrate drug combination; sacubitril; Valsartan; Ramipril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LCZ696 (sacubitril/valsartan) (Experimental): Following randomization, patients will receive LCZ696 in titrated doses from level 1 up to level 3 (50, 100 and 200 mg twice daily).
  Patients will be required to take a total of two pills, (one tablet from the LCZ696 pack and one capsule from ramipril matching placebo pack) twice a day for the duration of the study.
  Patients randomized to LCZ who were previously treated with ACE inhibitors receiving the last dose of that agent during the last 36 hours prior to randomization will receive a valsartan bridge for one day. These patients will receive two doses of valsartan for 1 day in a blinded manner prior to beginning double-blind LCZ696 treatment.
  Interventions: Drug: LCZ696 (sacubitril/valsartan); Drug: Placebo of ramipril; Drug: Valsartan
- Ramipril (Active Comparator): Following randomization, patients will receive the Ramipril in titrated doses from level 1 up to level 3 (1.25, 2.5 and 5 mg twice daily).
  Patients will be required to take a total of two pills, (one capsule from the ramipril pack and one tablet from LCZ696 matching placebo pack) twice a day for the duration of the study.
  Patients randomized to ramipril who were previously treated with ACE inhibitors receiving the last dose of that agent during the last 36 hours prior to randomization will immediately start on double-blind ramipril; however, to maintain double blind/double dummy of the valsartan bridge, these patients will receive two doses of matching valsartan placebo for 1 day in a blinded manner prior to beginning double-blind LCZ696 placebo.
  Interventions: Drug: Ramipril; Drug: Placebo of LCZ696; Drug: Placebo of valsartan

INTERVENTIONS:
Drug: LCZ696 (sacubitril/valsartan) — LCZ696 (sacubitril/valsartan) tablet will be available in 24/26 mg, 49/51 mg and 97/103 mg, respectively
  Arms: LCZ696 (sacubitril/valsartan)
Drug: Ramipril — Ramipril 1.25 mg, 2.5 mg, and 5 mg oral capsules
  Arms: Ramipril
Drug: Placebo of LCZ696 — Matching placebo of LCZ696 tablets
  Arms: Ramipril
Drug: Placebo of ramipril — Matching placebo of ramipril capsule
  Arms: LCZ696 (sacubitril/valsartan)
Drug: Valsartan — Valsartan (VAL489) 40 mg and 80 mg tablets, two doses for 1 day to patients who were previously treated with ACE inhibitors receiving the last dose of that agent during the last 36 hours prior to randomization
  Arms: LCZ696 (sacubitril/valsartan)
Drug: Placebo of valsartan — matching placebo of valsartan for one day to patients who will be randomized to received ramipril
  Arms: Ramipril

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of LCZ696 titrated to a target dose of 200 mg twice daily, compared to ramipril titrated to a target dose of 5 mg twice daily.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of LCZ696 titrated to a target dose of 200 mg twice daily, compared to ramipril titrated to a target dose of 5 mg twice daily, in addition to conventional post-AMI treatment, in reducing the occurrence of composite endpoint of CV death, HF hospitalization and outpatient HF (time-to-first event analysis) in post-AMI patients with evidence of LV systolic dysfunction and/or pulmonary congestion, with no known prior history of chronic HF.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age.
2. Diagnosis of spontaneous AMI based on the universal MI definition* with randomization to occur between 12 hours and 7 days after index event presentation. (*patients with spontaneous MI event determined to be secondary to another medical condition such as anemia, hypotension, or arrhythmia OR thought to be caused by coronary vasospasm with document normal coronary arteries are not eligible; patients with clinical presentation thought to be related to Takotsubo cardiomyopathy are also not eligible)
3. Evidence of LV systolic dysfunction and/or pulmonary congestion requiring intravenous treatment associated with the index MI event defined as:

   * LVEF ≤40% after index MI presentation and prior to randomization and/or
   * Pulmonary congestion requiring intravenous treatment with diuretics, vasodilators, vasopressors and/or inotropes, during the index hospitalization
4. At least one of the following 8 risk factors:

   * Age ≥ 70 years
   * eGFR <60 mL/min/1.73 m^2 based on MDRD formula at screening visit
   * Type I or II diabetes mellitus
   * Documented history of prior MI
   * Atrial fibrillation as noted by ECG, associated with index MI
   * LVEF <30% associated with index MI
   * Worst Killip class III or IV associated with index MI requiring intravenous treatment
   * STEMI without reperfusion therapy within the first 24 hours after presentation
5. Hemodynamically stable defined as:

   * SBP ≥ 100 mmHg at randomization for patients who received ACEi/ARB during the last 24 hours prior to randomization
   * SBP ≥ 110 mmHg at randomization for patients who did not receive ACEi/ARB during the last 24 hours prior to randomization
   * No IV treatment with diuretics, vasodilators, vasopressors and/or inotropes during the 24 hours prior to randomization

Key Exclusion Criteria:

1. Known history of chronic HF prior to randomization
2. Cardiogenic shock within the last 24 hours prior to randomization
3. Persistent clinical HF at the time of randomization
4. Coronary artery bypass graft (CABG) performed or planned for index MI
5. Clinically significant right ventricular MI as index MI
6. Symptomatic hypotension at screening or randomization
7. Patients with a known history of angioedema
8. Stroke or transient ischemic attack within one month prior to randomization
9. Known or suspected bilateral renal artery stenosis
10. Clinically significant obstructive cardiomyopathy
11. Open-heart surgery performed within one month prior to randomization or planned cardiac surgery w/in the 3 months prior to randomization
12. eGFR < 30 ml/min/1.73 m^2 as measured by MDRD at screening
13. Serum potassium > 5.2 mmol /L (or equivalent plasma potassium value) at randomization
14. Known hepatic impairment (as evidenced by total bilirubin > 3.0 mg/dL or increased ammonia levels, if performed), or history of cirrhosis with evidence of portal hypertension such as esophageal varices
15. Previous use of LCZ696
16. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin) within the past 3 years with a life expectancy of less than 1year.
17. History of hypersensitivity to the study drugs or drugs of similar chemical classes or known intolerance or contraindications to study drugs or drugs of similar chemical classes including ACE inhibitors, ARB or NEP inhibitors
18. Pregnant or nursing women or women of child-bearing potential unless they are using highly effective methods of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5669 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (421):
- United States (77):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Huntsville, Alabama
  - Novartis Investigative Site, Gilbert, Arizona
  - Novartis Investigative Site, Bakersfield, California
  - Novartis Investigative Site, Carmichael, California
  - Novartis Investigative Site, Los Alamitos, California
  - Novartis Investigative Site, Northridge, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Sylmar, California
  - Novartis Investigative Site, Brandon, Florida
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Jacksonville Beach, Florida
  - Novartis Investigative Site, Ocala, Florida
  - Novartis Investigative Site, Cumming, Georgia
  - Novartis Investigative Site, Johns Creek, Georgia
  - Novartis Investigative Site, Thomasville, Georgia
  - Novartis Investigative Site, Boise, Idaho
  - Novartis Investigative Site, Coeur d'Alene, Idaho
  - Novartis Investigative Site, Muncie, Indiana
  - Novartis Investigative Site, Munster, Indiana
  - Novartis Investigative Site, Richmond, Indiana
  - Novartis Investigative Site, Iowa City, Iowa
  - Novartis Investigative Site, Alexandria, Louisiana
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, Covington, Louisiana
  - Novartis Investigative Site, Hammond, Louisiana
  - Novartis Investigative Site, Slidell, Louisiana
  - Novartis Investigative Site, Bangor, Maine
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Rockville, Maryland
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Kalamazoo, Michigan
  - Novartis Investigative Site, Lansing, Michigan
  - Novartis Investigative Site, Petoskey, Michigan
  - Novartis Investigative Site, Saginaw, Michigan
  - Novartis Investigative Site, Southfield, Michigan
  - Novartis Investigative Site, Duluth, Minnesota
  - Novartis Investigative Site, Robbinsdale, Minnesota
  - Novartis Investigative Site, Saint Cloud, Minnesota
  - Novartis Investigative Site, Saint Paul, Minnesota
  - Novartis Investigative Site, Hattiesburg, Mississippi
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Lee's Summit, Missouri
  - Novartis Investigative Site, North Kansas City, Missouri
  - Novartis Investigative Site, Springfield, Missouri
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Lebanon, New Hampshire
  - Novartis Investigative Site, Hackensack, New Jersey
  - Novartis Investigative Site, Flushing, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Valhalla, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Grand Forks, North Dakota
  - Novartis Investigative Site, Canton, Ohio
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Erie, Pennsylvania
  - Novartis Investigative Site, Hershey, Pennsylvania
  - Novartis Investigative Site, York, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Rapid City, South Dakota
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Webster, Texas
  - Novartis Investigative Site, Danville, Virginia
  - Novartis Investigative Site, Falls Church, Virginia
  - Novartis Investigative Site, Lynchburg, Virginia
  - Novartis Investigative Site, Manassas, Virginia
  - Novartis Investigative Site, Bellevue, Washington
- Argentina (13):
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Buenos Aires, Buenos Aires F.D.
  - Novartis Investigative Site, Salta, Salta Province
  - Novartis Investigative Site, San Miguel de Tucumán, San Miguel de Tucuman
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Corrientes
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Formosa
  - Novartis Investigative Site, San Luis
  - Novartis Investigative Site, Santa Fe
- Australia (6):
  - Novartis Investigative Site, Chemside, Queensland
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, Bedford Park, South Australia
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, Geelong, Victoria
  - Novartis Investigative Site, Murdoch, Western Australia
- Austria (7):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Braunau am Inn
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Sankt Pölten
  - Novartis Investigative Site, Vienna
- Belgium (7):
  - Novartis Investigative Site, Edegem, Antwerpen
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Brasschaat
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Turnhout
  - Novartis Investigative Site, Yvoir
- Brazil (12):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Uberlândia, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Blumenau, Santa Catarina
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, São José do Rio Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Campina Grande do Sul
  - Novartis Investigative Site, São José
- Bulgaria (12):
  - Novartis Investigative Site, Burgas, BGR
  - Novartis Investigative Site, Sofia, BGR
  - Novartis Investigative Site, Blagoevgrad
  - Novartis Investigative Site, Burgas
  - Novartis Investigative Site, Gabrovo
  - Novartis Investigative Site, Kardzhali
  - Novartis Investigative Site, Pernik
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Rousse
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Canada (8):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
  - Novartis Investigative Site, Terrebonne, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- China (22):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Xicheng, Beijing Municipality
  - Novartis Investigative Site, Lanzhou, Gansu
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Yanji, Jilin
  - Novartis Investigative Site, Shengyang, Liaoning
  - Novartis Investigative Site, Jinan, Shandong
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Zhujing, Shanghai Municipality
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
  - Novartis Investigative Site, Wuhan
- Colombia (5):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Bucaramanga, Santander Department
  - Novartis Investigative Site, Cali, Valle del Cauca Department
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
- Croatia (3):
  - Novartis Investigative Site, Zagreb, HRV
  - Novartis Investigative Site, Čakovec
  - Novartis Investigative Site, Zagreb
- Czechia (6):
  - Novartis Investigative Site, Kladno, Czech Republic
  - Novartis Investigative Site, Liberec, Czech Republic
  - Novartis Investigative Site, Zlín, Czech Republic
  - Novartis Investigative Site, Brno-Bohunice
  - Novartis Investigative Site, Plzen-Bory
  - Novartis Investigative Site, Prague
- Denmark (7):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Glostrup Municipality
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Hvidovre
  - Novartis Investigative Site, Svendborg
  - Novartis Investigative Site, Vejle
  - Novartis Investigative Site, Viborg
- Finland (3):
  - Novartis Investigative Site, Jyväskylä
  - Novartis Investigative Site, Kaupio
  - Novartis Investigative Site, Tampere
- France (8):
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Chambray-lès-Tours
  - Novartis Investigative Site, Corbeil-Essonnes
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Toulouse
- Germany (30):
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Krozingen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Coburg
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Esslingen am Neckar
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Gütersloh
  - Novartis Investigative Site, Hennigsdorf
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Koeln-Nippes
  - Novartis Investigative Site, Langen
  - Novartis Investigative Site, Leverkusen
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Mönchengladbach
  - Novartis Investigative Site, Neuss
  - Novartis Investigative Site, Neuwied
  - Novartis Investigative Site, Riesa
  - Novartis Investigative Site, Rüsselsheim am Main
  - Novartis Investigative Site, Stadtlohn
  - Novartis Investigative Site, Vechta
  - Novartis Investigative Site, Villingen-Schwenningen
  - Novartis Investigative Site, Witten
  - Novartis Investigative Site, Würzburg
- Greece (4):
  - Novartis Investigative Site, Alexandroupoli, Evros
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Larissa, GR
  - Novartis Investigative Site, Athens
- Hungary (6):
  - Novartis Investigative Site, Pécs, Baranya
  - Novartis Investigative Site, Zalaegerszeg, Zala County
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Székesfehérvár
- India (15):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Karamsad, Gujarat
  - Novartis Investigative Site, Vadodara, Gujarat
  - Novartis Investigative Site, Gurgaon, Haryana
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Bikaner, Rajasthan
  - Novartis Investigative Site, Madurai, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Secunderabad, Telangana
  - Novartis Investigative Site, Dehradun, Uttarakhand
- Israel (6):
  - Novartis Investigative Site, Lower Galilee, Israel
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Sefad
  - Novartis Investigative Site, Tel Aviv
- Italy (13):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Catanzaro, CZ
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Grosseto, GR
  - Novartis Investigative Site, Sanremo, IM
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Rimini, RN
  - Novartis Investigative Site, Trieste, TS
  - Novartis Investigative Site, Napoli
- Mexico (6):
  - Novartis Investigative Site, Torreón, Coahulia
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Culiacan Sinaloa, Mexico City
  - Novartis Investigative Site, Mexico City
  - Novartis Investigative Site, Querétaro
  - Novartis Investigative Site, San Luis Potosí City
- Netherlands (20):
  - Novartis Investigative Site, Sneek, The Netherlands
  - Novartis Investigative Site, Alkmaar
  - Novartis Investigative Site, Almelo
  - Novartis Investigative Site, Amersfoort
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Beverwijk
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Ede
  - Novartis Investigative Site, Gouda
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Heemstede
  - Novartis Investigative Site, Leeuwarden
  - Novartis Investigative Site, Leiderdorp
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Tilburg
  - Novartis Investigative Site, Uden
  - Novartis Investigative Site, Veldhoven
  - Novartis Investigative Site, Venlo
  - Novartis Investigative Site, Zutphen
  - Novartis Investigative Site, Zwolle
- Norway (3):
  - Novartis Investigative Site, Grålum
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Stavanger
- Peru (4):
  - Novartis Investigative Site, Bellavista, Lima region
  - Novartis Investigative Site, Jesus Maria, Lima region
  - Novartis Investigative Site, Lima Cercado, Lima region
  - Novartis Investigative Site, Lima
- Philippines (3):
  - Novartis Investigative Site, Iloilo City, Iloilo
  - Novartis Investigative Site, Quezon City, Manila
  - Novartis Investigative Site, Manila, National Capital Region
- Poland (4):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Lubin
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Warsaw
- Portugal (10):
  - Novartis Investigative Site, Carnaxide, Lisbon District
  - Novartis Investigative Site, Almada
  - Novartis Investigative Site, Braga
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Covilha
  - Novartis Investigative Site, Faro
  - Novartis Investigative Site, Guimarães
  - Novartis Investigative Site, Leiria
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Vila Real
- Romania (14):
  - Novartis Investigative Site, Piteşti, Argeş
  - Novartis Investigative Site, Bucharest, District 4
  - Novartis Investigative Site, Oradea, Jud Bihor
  - Novartis Investigative Site, Cluj-Napoca, Jud Cluj
  - Novartis Investigative Site, Iași, Jud Iasi
  - Novartis Investigative Site, Târgu Mureş, Mureș County
  - Novartis Investigative Site, Brăila, ROM
  - Novartis Investigative Site, Suceava, ROM
  - Novartis Investigative Site, Timișoara, Timiș County
  - Novartis Investigative Site, Baia Mare
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Craiova
  - Novartis Investigative Site, Sibiu
  - Novartis Investigative Site, Timișoara
- Russia (15):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Murmansk
  - Novartis Investigative Site, N.Novgorod
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, S.-Petersburg
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Sestroretsk
  - Novartis Investigative Site, Sochy
  - Novartis Investigative Site, Tomsk
  - Novartis Investigative Site, Yekaterinburg
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (6):
  - Novartis Investigative Site, Bratislava, Slovak Republic
  - Novartis Investigative Site, Nitra, Slovak Republic
  - Novartis Investigative Site, Banská Bystrica, SVK
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Prešov
- South Africa (5):
  - Novartis Investigative Site, Pinelands, Cape Town
  - Novartis Investigative Site, Cape Town, Western Cape
  - Novartis Investigative Site, George, Western Cape
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Worcester
- South Korea (4):
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Cheongju-si, North Chungcheong
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Seoul
- Spain (12):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Villamartín, Cadiz
  - Novartis Investigative Site, León, Castille and León
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Cáceres, Extremadura
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Sweden (7):
  - Novartis Investigative Site, Stockholm, SE
  - Novartis Investigative Site, Goethenburg
  - Novartis Investigative Site, Helsingborg
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
  - Novartis Investigative Site, Västerås
- Switzerland (4):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lucerne
  - Novartis Investigative Site, Lugano
  - Novartis Investigative Site, Sankt Gallen
- Taiwan (6):
  - Novartis Investigative Site, New Taipei City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
  - Novartis Investigative Site, Yilan
- Thailand (4):
  - Novartis Investigative Site, Bangkok, THA
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Turkey (Türkiye) (9):
  - Novartis Investigative Site, Meselik, Eskişehir
  - Novartis Investigative Site, Ankara-Cankaya
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Kucukcekmece Istanbul
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Sivas
  - Novartis Investigative Site, Trabzon
- United Kingdom (14):
  - Novartis Investigative Site, Basingstoke, Hampshire
  - Novartis Investigative Site, Lincoln, Lincolnshire
  - Novartis Investigative Site, Craigavon, Northern Ireland
  - Novartis Investigative Site, Clydebank, West Dumbartonshire
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Bournemouth
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Middlesbrough
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Norwich
  - Novartis Investigative Site, Worcester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Curtain JP, Pfeffer MA, Braunwald E, Claggett BL, Granger CB, Kober L, Lewis EF, Maggioni AP, Mann DL, Rouleau JL, Solomon SD, Steg PG, Finn PV, Fernandez A, Jering KS, McMurray JJV. Rates of Sudden Death After Myocardial Infarction-Insights From the VALIANT and PARADISE-MI Trials. JAMA Cardiol. 2024 Oct 1;9(10):928-933. doi: 10.1001/jamacardio.2024.2356. PMID 39110471
- [Derived] Mann DL, Nicolas J, Claggett B, Miao ZM, Granger CB, Kerkar P, Kober L, Lewis EF, McMurray JJV, Maggioni AP, Nunez J, Ntsekhe M, Rouleau JL, Sim D, Solomon SD, Steg PG, van der Meer P, Braunwald E, Pfeffer MA, Mehran R. Angiotensin Receptor-Neprilysin Inhibition in Patients With STEMI vs NSTEMI. J Am Coll Cardiol. 2024 Mar 5;83(9):904-914. doi: 10.1016/j.jacc.2024.01.002. PMID 38418004
- [Derived] Petrie MC, Rouleau JL, Claggett B, Jering K, van der Meer P, Kober L, Miao ZM, Lewis E, Granger C, De Pasqulae CG, Mann D, Steg PG, Maggioni A, Amir O, Lefkowitz M, Braunwald E, Solomon SD, McMurray JJV, Pfeffer MA. Pulmonary Congestion and Left Ventricular Dysfunction After Myocardial Infarction: Insights From the PARADISE-MI Trial. Circulation. 2024 Jan 23;149(4):335-338. doi: 10.1161/CIRCULATIONAHA.123.066163. Epub 2024 Jan 22. No abstract available. PMID 38252738
- [Derived] Wang X, Jering KS, Cikes M, Tokmakova MP, Mehran R, Han Y, East C, Mody FV, Wang Y, Lewis EF, Claggett B, McMurray JJV, Granger CB, Pfeffer MA, Solomon SD. Sex Differences in Clinical Characteristics and Outcomes After Myocardial Infarction With Low Ejection Fraction: Insights From PARADISE-MI. J Am Heart Assoc. 2023 Sep 5;12(17):e028942. doi: 10.1161/JAHA.122.028942. Epub 2023 Aug 23. PMID 37609931
- [Derived] Jering KS, Claggett BL, Pfeffer MA, Granger CB, Kober L, Lewis EF, Maggioni AP, Mann DL, McMurray JJV, Prescott MF, Rouleau JL, Solomon SD, Steg PG, von Lewinski D, Braunwald E. Prognostic Importance of NT-proBNP (N-Terminal Pro-B-Type Natriuretic Peptide) Following High-Risk Myocardial Infarction in the PARADISE-MI Trial. Circ Heart Fail. 2023 May;16(5):e010259. doi: 10.1161/CIRCHEARTFAILURE.122.010259. Epub 2023 May 1. PMID 37125529
- [Derived] Mehran R, Steg PG, Pfeffer MA, Jering K, Claggett B, Lewis EF, Granger C, Kober L, Maggioni A, Mann DL, McMurray JJV, Rouleau JL, Solomon SD, Ducrocq G, Berwanger O, De Pasquale CG, Landmesser U, Petrie M, Leng DSK, van der Meer P, Lefkowitz M, Zhou Y, Braunwald E. The Effects of Angiotensin Receptor-Neprilysin Inhibition on Major Coronary Events in Patients With Acute Myocardial Infarction: Insights From the PARADISE-MI Trial. Circulation. 2022 Dec 6;146(23):1749-1757. doi: 10.1161/CIRCULATIONAHA.122.060841. Epub 2022 Nov 2. PMID 36321459
- [Derived] Shah AM, Claggett B, Prasad N, Li G, Volquez M, Jering K, Cikes M, Kovacs A, Mullens W, Nicolau JC, Kober L, van der Meer P, Jhund PS, Ibram G, Lefkowitz M, Zhou Y, Solomon SD, Pfeffer MA. Impact of Sacubitril/Valsartan Compared With Ramipril on Cardiac Structure and Function After Acute Myocardial Infarction: The PARADISE-MI Echocardiographic Substudy. Circulation. 2022 Oct 4;146(14):1067-1081. doi: 10.1161/CIRCULATIONAHA.122.059210. Epub 2022 Sep 9. PMID 36082663
- [Derived] Pfeffer MA, Claggett B, Lewis EF, Granger CB, Kober L, Maggioni AP, Mann DL, McMurray JJV, Rouleau JL, Solomon SD, Steg PG, Berwanger O, Cikes M, De Pasquale CG, Fernandez A, Filippatos G, Jering K, Landmesser U, Menon V, Merkely B, Petrie MC, Petrov I, Schou M, Senni M, Sim D, van der Meer P, Lefkowitz M, Zhou Y, Wang Y, Braunwald E. Impact of Sacubitril/Valsartan Versus Ramipril on Total Heart Failure Events in the PARADISE-MI Trial. Circulation. 2022 Jan 4;145(1):87-89. doi: 10.1161/CIRCULATIONAHA.121.057429. Epub 2021 Nov 19. No abstract available. PMID 34797725
- [Derived] Pfeffer MA, Claggett B, Lewis EF, Granger CB, Kober L, Maggioni AP, Mann DL, McMurray JJV, Rouleau JL, Solomon SD, Steg PG, Berwanger O, Cikes M, De Pasquale CG, East C, Fernandez A, Jering K, Landmesser U, Mehran R, Merkely B, Vaghaiwalla Mody F, Petrie MC, Petrov I, Schou M, Senni M, Sim D, van der Meer P, Lefkowitz M, Zhou Y, Gong J, Braunwald E; PARADISE-MI Investigators and Committees. Angiotensin Receptor-Neprilysin Inhibition in Acute Myocardial Infarction. N Engl J Med. 2021 Nov 11;385(20):1845-1855. doi: 10.1056/NEJMoa2104508. PMID 34758252

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 5669 patients were randomized in a 1:1 ratio to the sacubitril/valsartan treatment group and the ramipril treatment group at 493 sites in 41 countries. A total of 8 patients were mis-randomized, 4 from each treatment group. One of the mis-randomized patients of the ramipril group died. The Full analysis set (FAS) was comprised of 5661 patients.
Groups:
- LCZ696 (Sacubitril/Valsartan): Following randomization, patients received LCZ696 in titrated doses from level 1 up to level 3 (50, 100 and 200 mg twice daily).
  Patients were required to take a total of two pills, (one tablet from the LCZ696 pack and one capsule from Ramipril matching placebo pack) twice a day for the duration of the study.
  Patients randomized to LCZ who were previously treated with ACE inhibitors, receiving the last dose of that agent during the last 36 hours prior to randomization, received a valsartan bridge for one day. These patients received two doses of valsartan for 1 day in a blinded manner prior to beginning double-blind LCZ696 treatment.
- Ramipril: Following randomization, patients received Ramipril in titrated doses from level 1 up to level 3 (1.25, 2.5 and 5 mg twice daily).
  Patients were required to take a total of two pills, (one capsule from the Ramipril pack and one tablet from LCZ696 matching placebo pack) twice a day for the duration of the study.
  Patients randomized to Ramipril who were previously treated with ACE inhibitors, receiving the last dose of that agent during the last 36 hours prior to randomization immediately started on double-blind ramipril; however, to maintain double blind/double dummy of the valsartan bridge, these patients received two doses of matching valsartan placebo for 1 day in a blinded manner prior to beginning double-blind LCZ696 placebo.
Period: Overall Study
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Ramipril
Started (All randomized patients (RAN)) | 2834 | 2835
Full Analysis Set (FAS) (All patients in the RAN population who were not mis-randomized patients (who were not qualified for randomization and who did not take study drug, but were inadvertently randomized into the study).) | 2830 | 2831
Safety Set (SAF) (All randomized patients who received at least one dose of study drug.) | 2820 | 2816
Completed | 2605 | 2576
Not Completed | 229 | 259
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Lost to Follow-up | 2 | 5
Not completed — Death | 221 | 247
Not completed — Mis-randomized (one mis-randomized patient in the Ramipril group also died) | 4 | 3

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of 5661 patients and consisted of patients in the Randomized population who were not mis-randomized patients. Out of the 5669 patients randomized, a total of 8 patients were mis-randomized, 4 from each treatment group. Following the intent-to-treat (ITT) principle, patients in the FAS were analyzed according to the treatment they were assigned to at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Ramipril | Total
Number analyzed (Participants) | 2830 | 2831 | 5661
Age, Customized [Count of Participants; unit: Participants] — Participants in age categories can be counted more than once in the appropriate category.
  Participants
    <65 years | 1386 | 1451 | 2837
    ≥65 years | 1444 | 1380 | 2824
    <75 years | 2286 | 2324 | 4610
    ≥75 years | 544 | 507 | 1051
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 663 | 700 | 1363
  Male | 2167 | 2131 | 4298
Race/Ethnicity, Customized [Number; unit: Participants] — Race/Ethnicity
  Participants
    Caucasian | 2125 | 2138 | 4263
    Black | 35 | 40 | 75
    Asian | 475 | 478 | 953
    Native American | 45 | 45 | 90
    Pacific Islander | 0 | 4 | 4
    Unknown | 22 | 21 | 43
    Other | 128 | 105 | 233

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First CEC (Clinical Endpoint Committee) Confirmed Primary Composite Endpoint
Description: A confirmed composite endpoint includes cardiovascular (CV) death, heart failure (HF) hospitalization, or outpatient heart failure
Time Frame: From randomization to first occurrence (up to approximately 43 months)
Population: Full Analysis Set
Measure: Number; unit: Count of Participants
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Ramipril
Number analyzed (Participants) | 2830 | 2831
Count of Participants
  Primary Composite | 338 | 373
  Cardiovascular (CV) Death | 168 | 191
  First Heart Failure (HF) Hospitalization | 170 | 195
  First Outpatient Heart Failure (HF) | 39 | 57
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Ramipril; Primary Composite; Test type: Superiority; p = 0.1659, Cox's Proportional Hazard Model; Hazard Ratio (HR) = 0.9012, 95% CI 2-sided [0.7778 to 1.0441]
Statistical Analysis 2: Comparison: LCZ696 (Sacubitril/Valsartan) vs Ramipril; CV Death; Test type: Superiority; p = 0.2031, Cox's Proportional Hazard Model; Hazard Ratio (HR) = 0.8740, 95% CI 2-sided [0.7104 to 1.0754]
Statistical Analysis 3: Comparison: LCZ696 (Sacubitril/Valsartan) vs Ramipril; First HF Hospitalization; Test type: Superiority; p = 0.1679, Cox's Proportional Hazard Model; Hazard Ratio (HR) = 0.8653, 95% CI 2-sided [0.7044 to 1.0629]
Statistical Analysis 4: Comparison: LCZ696 (Sacubitril/Valsartan) vs Ramipril; First Outpatient HF; Test type: Superiority; p = 0.0667, Cox's Proportional Hazard Model; Hazard Ratio (HR) = 0.6831, 95% CI 2-sided [0.4546 to 1.0266]

2. Secondary Outcome: Number of Participants With a Confirmed Composite of CV Death or HF Hospitalization
Description: A confirmed composite endpoint for this outcome measure includes cardiovascular death or heart failure hospitalization.
Time Frame: Time from randomization to first occurrence (up to approximately 43 months)
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Ramipril
Number analyzed (Participants) | 2830 | 2831
Participants | 308 | 335
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Ramipril; CV death or HF hospitalization; Test type: Superiority; p = 0.2507, Cox's Proportional Hazard Model; Hazard Ratio (HR) = 0.9133, 95% CI 2-sided [0.7824 to 1.0662]

3. Secondary Outcome: Number of Participants With a Confirmed Composite of HF Hospitalization or Outpatient HF
Description: A confirmed composite endpoint includes first occurrence of heart failure hospitalization or outpatient heart failure
Time Frame: Time from randomization to first occurrence (approximately up to 43 months)
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Ramipril
Number analyzed (Participants) | 2830 | 2831
Participants | 201 | 237
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Ramipril; HF hospitalization or Outpatient HF; Test type: Superiority; p = 0.0732, Cox's Proportional Hazard Model; Hazard Ratio (HR) = 0.8422, 95% CI 2-sided [0.6979 to 1.0163]

4. Secondary Outcome: Number of Participants With a Confirmed Composite of CV Death, Non-fatal Spontaneous Myocardial Infarction or Non-fatal Stroke
Description: A confirmed composite endpoint for this outcome measure includes cardiovascular death, non-fatal spontaneous myocardial infarction or non-fatal stroke
Time Frame: Time from randomization to first occurrence (approximately up to 43 months)
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Ramipril
Number analyzed (Participants) | 2830 | 2831
Participants | 315 | 349
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Ramipril; CV death, Non-fatal spontaneous MI or Non-fatal stroke; Test type: Superiority; p = 0.1785, Cox's Proportional Hazard Model; Hazard Ratio (HR) = 0.9007, 95% CI 2-sided [0.7734 to 1.0489]

5. Secondary Outcome: Total Number of Confirmed Composite Endpoints
Description: A confirmed composite endpoint includes cardiovascular death, heart failure hospitalization, non-fatal spontaneous MI hospitalization, and non-fatal stroke hospitalization
Time Frame: Time from randomization to end of study (approximately up to 43 months)
Population: Full Analysis Set
Measure: Number; unit: Events
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Ramipril
Number analyzed (Participants) | 2830 | 2831
Events | 416 | 455
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Ramipril; Total Number of Confirmed Composite Endpoints; Test type: Superiority; p = 0.0452, Negative Binomial regression model; Rate Ratio = 0.8361, 95% CI 2-sided [0.7018 to 0.9961]

6. Secondary Outcome: All-cause Mortality for Full Analysis Set (FAS)
Description: All-cause mortality defined as deaths related to Cardiovascular (CV) and non-CV events for patients in the Full Analysis Set up to a cut-off date of 31-Dec-2020.
Time Frame: Time from randomization to death (approximately up to 43 months)
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Ramipril
Number analyzed (Participants) | 2830 | 2831
Participants | 213 | 242
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Ramipril; All-Cause Death; Test type: Superiority; p = 0.1556, Cox's Proportional Hazard Model; Hazard Ratio (HR) = 0.8751, 95% CI 2-sided [0.7279 to 1.0520]

7. Post Hoc Outcome: All Collected Deaths
Description: Pre-treatment deaths were collected from randomization to the day before first dose of study medication, for a maximum duration of 5 days.
  On-treatment and post-treatment safety follow-up deaths were collected from first dose of study medication to 30 days after the last dose of study medication.
  All deaths refer to the sum of pre-treatment, on-treatment and post-treatment safety follow-up deaths.
Time Frame: Pre-treatment: Up to 5 days before Day 1. On-treatment and post-treatment safety follow up: up to 4 years
Population: All subjects to whom study treatment was assigned by randomization, regardless of whether or not treatment was administered
Measure: Number; unit: Participants
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Ramipril
Number analyzed (Participants) | 2834 | 2835
Participants
  pre-treatment deaths | 1 | 3
  On-treatment deaths and extended safety follow-up: number analyzed (Participants) | 2820 | 2816
  On-treatment deaths and extended safety follow-up | 220 | 244
  All deaths | 221 | 247

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of approximately 4 years. All-Cause Mortality was collected from randomization until the end of study treatment plus 30 days post-treatment, up to a maximum duration of approximately 4 years.
Description: Adverse Event: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment.
  All-Cause Mortality is using the Randomized Set, including patients who were not treated.
Groups:
- LCZ696 Pre-treatment: Only for pre-treatment deaths that are not included in the safety set.
- Ramipril Pre-treatment: Only pre-treatment deaths that are not included in the safety set
- LCZ696: Following randomization, patients received LCZ696 in titrated doses from level 1 up to level 3 (50, 100 and 200 mg twice daily).
  Patients were required to take a total of two pills, (one tablet from the LCZ696 pack and one capsule from Ramipril matching placebo pack) twice a day for the duration of the study.
  Patients randomized to LCZ who were previously treated with ACE inhibitors, receiving the last dose of that agent during the last 36 hours prior to randomization, received a valsartan bridge for one day. These patients received two doses of valsartan for 1 day in a blinded manner prior to beginning double-blind LCZ696 treatment.
Arm/Group | LCZ696 Pre-treatment | Ramipril Pre-treatment | LCZ696 | Ramipril
All-Cause Mortality (participants affected / at risk) | 1/2834 | 3/2835 | 220/2820 | 244/2816
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 1146/2820 | 1126/2816
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 1769/2820 | 1770/2816
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 Pre-treatment (N=0) | Ramipril Pre-treatment (N=0) | LCZ696 (N=2820) | Ramipril (N=2816)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 30 | 23
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1
Hypocoagulable state (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 7 | 4
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 3
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 11 | 13
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 9 | 6
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 92 | 95
Adams-Stokes syndrome (Cardiac disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 59 | 84
Angina unstable (Cardiac disorders) | 0 | 0 | 65 | 76
Anginal equivalent (Cardiac disorders) | 0 | 0 | 1 | 0
Aortic valve disease (Cardiac disorders) | 0 | 0 | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 9 | 3
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 2 | 5
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 30 | 22
Atrial flutter (Cardiac disorders) | 0 | 0 | 6 | 7
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 5 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 2 | 4
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 2 | 2
Bradycardia (Cardiac disorders) | 0 | 0 | 6 | 4
Cardiac aneurysm (Cardiac disorders) | 0 | 0 | 1 | 2
Cardiac arrest (Cardiac disorders) | 0 | 0 | 24 | 31
Cardiac asthma (Cardiac disorders) | 0 | 0 | 2 | 3
Cardiac discomfort (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac disorder (Cardiac disorders) | 0 | 0 | 2 | 2
Cardiac failure (Cardiac disorders) | 0 | 0 | 149 | 183
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 28 | 22
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 12 | 8
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 27 | 37
Cardiac perforation (Cardiac disorders) | 0 | 0 | 0 | 2
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 6
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 0 | 4 | 8
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 7 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 17 | 12
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiovascular insufficiency (Cardiac disorders) | 0 | 0 | 1 | 2
Chronic left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 23 | 30
Coronary artery insufficiency (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 3 | 6
Coronary artery perforation (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1 | 4
Dressler's syndrome (Cardiac disorders) | 0 | 0 | 1 | 2
Endocarditis noninfective (Cardiac disorders) | 0 | 0 | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 0 | 1 | 3
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 6 | 10
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 3 | 3
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 3
Microvascular coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 5 | 4
Myocardial fibrosis (Cardiac disorders) | 0 | 0 | 2 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 51 | 44
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 9 | 9
Palpitations (Cardiac disorders) | 0 | 0 | 4 | 1
Papillary muscle disorder (Cardiac disorders) | 0 | 0 | 1 | 0
Paroxysmal atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 2 | 6
Pericardial haemorrhage (Cardiac disorders) | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 6 | 8
Pulseless electrical activity (Cardiac disorders) | 0 | 0 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 2
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 3 | 3
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 2 | 3
Tachycardia (Cardiac disorders) | 0 | 0 | 3 | 1
Ventricle rupture (Cardiac disorders) | 0 | 0 | 1 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 2 | 5
Ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 2 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 12 | 11
Ventricular remodelling (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 19 | 23
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 4 | 5
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Adrenal mass (Endocrine disorders) | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Arteriosclerotic retinopathy (Eye disorders) | 0 | 0 | 0 | 1
Blindness unilateral (Eye disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 3 | 2
Diplopia (Eye disorders) | 0 | 0 | 2 | 0
Eye oedema (Eye disorders) | 0 | 0 | 0 | 1
Eye swelling (Eye disorders) | 0 | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 1
Intraocular haematoma (Eye disorders) | 0 | 0 | 1 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 0 | 1
Open angle glaucoma (Eye disorders) | 0 | 0 | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0
Rhegmatogenous retinal detachment (Eye disorders) | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 2 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 8 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 7 | 5
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 4
Colitis (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dental cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 4 | 8
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 3 | 2
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 5
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 15 | 12
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 4 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 5 | 2
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Malabsorption (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 7 | 1
Mesenteric arterial occlusion (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mouth swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 5 | 1
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 2 | 5
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Peritoneal adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 3 | 6
Rectal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 3 | 3
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 5 | 5
Adverse event (General disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 3 | 3
Cardiac death (General disorders) | 0 | 0 | 5 | 4
Chest discomfort (General disorders) | 0 | 0 | 3 | 2
Chest pain (General disorders) | 0 | 0 | 1 | 2
Complication associated with device (General disorders) | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 27 | 31
Disease progression (General disorders) | 0 | 0 | 0 | 1
Drowning (General disorders) | 0 | 0 | 1 | 0
Exercise tolerance decreased (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 2
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 1 | 0
Hypothermia (General disorders) | 0 | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1 | 2
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 3 | 3
Necrosis (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 54 | 66
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Polyp (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 7 | 3
Sudden cardiac death (General disorders) | 0 | 0 | 10 | 14
Sudden death (General disorders) | 0 | 0 | 9 | 8
Surgical failure (General disorders) | 0 | 0 | 0 | 1
Ulcer haemorrhage (General disorders) | 0 | 0 | 0 | 1
Unevaluable event (General disorders) | 0 | 0 | 1 | 0
Vascular stent stenosis (General disorders) | 0 | 0 | 5 | 5
Vascular stent thrombosis (General disorders) | 0 | 0 | 7 | 7
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1 | 2
Biliary cyst (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Biliary dyspepsia (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 4 | 9
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 9 | 6
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 4 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic mass (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 2
Abscess (Infections and infestations) | 0 | 0 | 2 | 0
Abscess jaw (Infections and infestations) | 0 | 0 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 3 | 2
Abscess oral (Infections and infestations) | 0 | 0 | 1 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 2 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 3 | 3
Bacteraemia (Infections and infestations) | 0 | 0 | 3 | 1
Bacterial abdominal infection (Infections and infestations) | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Biliary sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Bone abscess (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 3 | 6
COVID-19 (Infections and infestations) | 0 | 0 | 13 | 16
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 6 | 8
Carbuncle (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 11 | 5
Cholangitis infective (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 4 | 3
Cystitis (Infections and infestations) | 0 | 0 | 7 | 2
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1
Diabetic foot infection (Infections and infestations) | 0 | 0 | 1 | 1
Diabetic gangrene (Infections and infestations) | 0 | 0 | 1 | 2
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 3 | 2
Empyema (Infections and infestations) | 0 | 0 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 3 | 0
Endocarditis staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0
Endometritis (Infections and infestations) | 0 | 0 | 1 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 6 | 5
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 2 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Fournier's gangrene (Infections and infestations) | 0 | 0 | 1 | 1
Gangrene (Infections and infestations) | 0 | 0 | 3 | 5
Gas gangrene (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 11 | 7
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 2
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 0 | 0 | 1
Helicobacter duodenal ulcer (Infections and infestations) | 0 | 0 | 1 | 0
Implant site infection (Infections and infestations) | 0 | 0 | 0 | 1
Incision site abscess (Infections and infestations) | 0 | 0 | 1 | 0
Infected dermal cyst (Infections and infestations) | 0 | 0 | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 4 | 3
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 3 | 2
Joint abscess (Infections and infestations) | 0 | 0 | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 1 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 4 | 2
Lung abscess (Infections and infestations) | 0 | 0 | 1 | 0
Meningitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Orchitis (Infections and infestations) | 0 | 0 | 1 | 2
Osteomyelitis (Infections and infestations) | 0 | 0 | 4 | 1
Osteomyelitis acute (Infections and infestations) | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0
Parotitis (Infections and infestations) | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 3
Pharyngeal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 61 | 73
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 3 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 0 | 1 | 0
Post procedural sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 3
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 2 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 3 | 2
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 3 | 1
Pyelonephritis chronic (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 3 | 6
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 0 | 2 | 0
Scrotal abscess (Infections and infestations) | 0 | 0 | 2 | 0
Sepsis (Infections and infestations) | 0 | 0 | 19 | 13
Septic shock (Infections and infestations) | 0 | 0 | 9 | 8
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 2
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 2 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 28 | 16
Urosepsis (Infections and infestations) | 0 | 0 | 6 | 2
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 1 | 0
Viral labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 1
Viral sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Wound abscess (Infections and infestations) | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 3
Wound infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Accidental exposure to product (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Anastomotic leak (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | NA | NA | 3 | 2
Arterial bypass occlusion (Injury, poisoning and procedural complications) | NA | NA | 2 | 0
Arterial injury (Injury, poisoning and procedural complications) | NA | NA | 3 | 1
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Cardiac procedure complication (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Cardiac valve rupture (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Concussion (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Contusion (Injury, poisoning and procedural complications) | NA | NA | 4 | 5
Coronary artery restenosis (Injury, poisoning and procedural complications) | NA | NA | 0 | 3
Coronary bypass thrombosis (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Coronary vascular graft occlusion (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | NA | NA | 1 | 2
Electric shock (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Fall (Injury, poisoning and procedural complications) | NA | NA | 5 | 7
Femoral neck fracture (Injury, poisoning and procedural complications) | NA | NA | 2 | 1
Femur fracture (Injury, poisoning and procedural complications) | NA | NA | 4 | 4
Fibula fracture (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | NA | NA | 1 | 1
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Fracture (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Head injury (Injury, poisoning and procedural complications) | NA | NA | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | NA | NA | 2 | 3
Humerus fracture (Injury, poisoning and procedural complications) | NA | NA | 2 | 0
Incisional hernia (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | NA | NA | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | NA | NA | 0 | 3
Limb injury (Injury, poisoning and procedural complications) | NA | NA | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | NA | NA | 1 | 1
Muscle injury (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | NA | NA | 0 | 2
Overdose (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Periorbital haemorrhage (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | NA | NA | 2 | 2
Pneumothorax traumatic (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Poisoning (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Post intensive care syndrome (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | NA | NA | 1 | 3
Post procedural discharge (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | NA | NA | 4 | 2
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Post procedural urine leak (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Prevertebral soft tissue swelling of cervical space (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Pulmonary contusion (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | NA | NA | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | NA | NA | 1 | 3
Road traffic accident (Injury, poisoning and procedural complications) | NA | NA | 0 | 2
Skin abrasion (Injury, poisoning and procedural complications) | NA | NA | 1 | 2
Skin laceration (Injury, poisoning and procedural complications) | NA | NA | 1 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Stomal hernia (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | NA | NA | 1 | 4
Subdural haemorrhage (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | NA | NA | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | NA | NA | 3 | 3
Vasoplegia syndrome (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | NA | NA | 0 | 2
Wrist fracture (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Angiocardiogram (Investigations) | NA | NA | 2 | 1
Anticoagulation drug level above therapeutic (Investigations) | NA | NA | 1 | 0
Biopsy bladder (Investigations) | NA | NA | 1 | 0
Biopsy prostate (Investigations) | NA | NA | 1 | 0
Blood creatinine increased (Investigations) | NA | NA | 0 | 2
Blood glucose fluctuation (Investigations) | NA | NA | 0 | 1
Blood glucose increased (Investigations) | NA | NA | 2 | 0
Blood sodium decreased (Investigations) | NA | NA | 0 | 1
Cardiac output decreased (Investigations) | NA | NA | 1 | 0
Cardiac ventriculogram (Investigations) | NA | NA | 0 | 1
Coagulation test abnormal (Investigations) | NA | NA | 0 | 1
Ejection fraction (Investigations) | NA | NA | 1 | 1
Ejection fraction abnormal (Investigations) | NA | NA | 0 | 1
Ejection fraction decreased (Investigations) | NA | NA | 6 | 12
Electrocardiogram QT prolonged (Investigations) | NA | NA | 1 | 0
Glycosylated haemoglobin increased (Investigations) | NA | NA | 0 | 1
Haemoglobin decreased (Investigations) | NA | NA | 2 | 0
Heart rate decreased (Investigations) | NA | NA | 0 | 1
Hepatic enzyme increased (Investigations) | NA | NA | 0 | 1
Influenza B virus test positive (Investigations) | NA | NA | 0 | 1
International normalised ratio increased (Investigations) | NA | NA | 1 | 0
Liver function test abnormal (Investigations) | NA | NA | 0 | 2
Liver function test increased (Investigations) | NA | NA | 1 | 0
Neutrophil count decreased (Investigations) | NA | NA | 0 | 1
Occult blood positive (Investigations) | NA | NA | 1 | 0
Renal function test abnormal (Investigations) | NA | NA | 1 | 0
SARS-CoV-2 test positive (Investigations) | NA | NA | 1 | 2
Scan myocardial perfusion abnormal (Investigations) | NA | NA | 1 | 0
Stress echocardiogram (Investigations) | NA | NA | 0 | 1
Transaminases increased (Investigations) | NA | NA | 1 | 0
Troponin increased (Investigations) | NA | NA | 1 | 0
Weight decreased (Investigations) | NA | NA | 1 | 1
Weight increased (Investigations) | NA | NA | 1 | 1
Acidosis hyperchloraemic (Metabolism and nutrition disorders) | NA | NA | 0 | 1
Cachexia (Metabolism and nutrition disorders) | NA | NA | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | NA | NA | 1 | 2
Dehydration (Metabolism and nutrition disorders) | NA | NA | 9 | 10
Diabetes mellitus (Metabolism and nutrition disorders) | NA | NA | 2 | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | NA | NA | 1 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | NA | NA | 3 | 2
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | NA | NA | 2 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | NA | NA | 1 | 0
Euglycaemic diabetic ketoacidosis (Metabolism and nutrition disorders) | NA | NA | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | NA | NA | 2 | 2
Food intolerance (Metabolism and nutrition disorders) | NA | NA | 1 | 0
Gout (Metabolism and nutrition disorders) | NA | NA | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | NA | NA | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | NA | NA | 6 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | NA | NA | 15 | 4
Hypertriglyceridaemia (Metabolism and nutrition disorders) | NA | NA | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | NA | NA | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | NA | NA | 7 | 10
Hypokalaemia (Metabolism and nutrition disorders) | NA | NA | 5 | 3
Hyponatraemia (Metabolism and nutrition disorders) | NA | NA | 3 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | NA | NA | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | NA | NA | 1 | 1
Ketoacidosis (Metabolism and nutrition disorders) | NA | NA | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | NA | NA | 0 | 2
Malnutrition (Metabolism and nutrition disorders) | NA | NA | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | NA | NA | 2 | 1
Obesity (Metabolism and nutrition disorders) | NA | NA | 1 | 1
Pseudohyponatraemia (Metabolism and nutrition disorders) | NA | NA | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | NA | NA | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | NA | NA | 4 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | NA | NA | 1 | 2
Arthritis reactive (Musculoskeletal and connective tissue disorders) | NA | NA | 0 | 1
Back disorder (Musculoskeletal and connective tissue disorders) | NA | NA | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | NA | NA | 2 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | NA | NA | 0 | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | NA | NA | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | NA | NA | 2 | 0
Deformity thorax (Musculoskeletal and connective tissue disorders) | NA | NA | 1 | 0
Enthesopathy (Musculoskeletal and connective tissue disorders) | NA | NA | 0 | 1
Fistula discharge (Musculoskeletal and connective tissue disorders) | NA | NA | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | NA | NA | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | NA | NA | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | NA | NA | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | NA | NA | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | NA | NA | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | NA | NA | 2 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | NA | NA | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | NA | NA | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | NA | NA | 5 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | NA | NA | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | NA | NA | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | NA | NA | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | NA | NA | 3 | 6
Osteochondrosis (Musculoskeletal and connective tissue disorders) | NA | NA | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | NA | NA | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | NA | NA | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | NA | NA | 1 | 0
Periostosis (Musculoskeletal and connective tissue disorders) | NA | NA | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | NA | NA | 1 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | NA | NA | 1 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | NA | NA | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | NA | NA | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | NA | NA | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 2
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Anaplastic meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
B-cell unclassifiable lymphoma low grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 4 | 3
Benign duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 4 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 2 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 2 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 3 | 1
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 2 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 5
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 2 | 1
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 3 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Gallbladder adenosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 1
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 1
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 2
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 2
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 2
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 2 | 5
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 3
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 2 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 2 | 1
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0
Myxoid liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 2
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 2
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 3 | 0
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 3 | 0
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0
Pleural mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 5 | 3
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 2 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 3 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 4 | 1
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 3
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 2 | 1
Squamous cell carcinoma of the parotid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 | 1
Arachnoid cyst (Nervous system disorders) | NA | NA | 0 | 1
Ataxia (Nervous system disorders) | NA | NA | 1 | 0
Brain stem ischaemia (Nervous system disorders) | NA | NA | 1 | 0
Carotid artery occlusion (Nervous system disorders) | NA | NA | 0 | 1
Carotid artery stenosis (Nervous system disorders) | NA | NA | 5 | 2
Cerebellar infarction (Nervous system disorders) | NA | NA | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | NA | NA | 1 | 1
Cerebral hypoperfusion (Nervous system disorders) | NA | NA | 1 | 0
Cerebral infarction (Nervous system disorders) | NA | NA | 8 | 9
Cerebral ischaemia (Nervous system disorders) | NA | NA | 2 | 0
Cerebral venous sinus thrombosis (Nervous system disorders) | NA | NA | 1 | 0
Cerebrovascular accident (Nervous system disorders) | NA | NA | 32 | 33
Cerebrovascular disorder (Nervous system disorders) | NA | NA | 1 | 0
Cerebrovascular insufficiency (Nervous system disorders) | NA | NA | 1 | 0
Cervical radiculopathy (Nervous system disorders) | NA | NA | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | NA | NA | 1 | 0
Demyelinating polyneuropathy (Nervous system disorders) | NA | NA | 1 | 1
Disturbance in attention (Nervous system disorders) | NA | NA | 0 | 1
Dizziness (Nervous system disorders) | NA | NA | 7 | 3
Dizziness postural (Nervous system disorders) | NA | NA | 1 | 1
Dysarthria (Nervous system disorders) | NA | NA | 1 | 2
Embolic stroke (Nervous system disorders) | NA | NA | 1 | 0
Encephalopathy (Nervous system disorders) | NA | NA | 0 | 2
Epilepsy (Nervous system disorders) | NA | NA | 0 | 2
Facial paralysis (Nervous system disorders) | NA | NA | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | NA | NA | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | NA | NA | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | NA | NA | 2 | 2
Haemorrhagic transformation stroke (Nervous system disorders) | NA | NA | 0 | 1
Headache (Nervous system disorders) | NA | NA | 2 | 2
Hemianopia (Nervous system disorders) | NA | NA | 1 | 0
Hemiparesis (Nervous system disorders) | NA | NA | 2 | 0
Hypoaesthesia (Nervous system disorders) | NA | NA | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | NA | NA | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | NA | NA | 2 | 0
Irregular sleep wake rhythm disorder (Nervous system disorders) | NA | NA | 1 | 0
Ischaemic stroke (Nervous system disorders) | NA | NA | 12 | 15
Lacunar infarction (Nervous system disorders) | NA | NA | 1 | 0
Lacunar stroke (Nervous system disorders) | NA | NA | 0 | 1
Loss of consciousness (Nervous system disorders) | NA | NA | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | NA | NA | 2 | 1
Migraine (Nervous system disorders) | NA | NA | 0 | 1
Moyamoya disease (Nervous system disorders) | NA | NA | 0 | 1
Neuropathy peripheral (Nervous system disorders) | NA | NA | 0 | 1
Paraesthesia (Nervous system disorders) | NA | NA | 1 | 0
Partial seizures (Nervous system disorders) | NA | NA | 0 | 1
Polyneuropathy (Nervous system disorders) | NA | NA | 1 | 0
Post stroke seizure (Nervous system disorders) | NA | NA | 0 | 1
Presyncope (Nervous system disorders) | NA | NA | 9 | 4
Psychogenic seizure (Nervous system disorders) | NA | NA | 1 | 0
Radiculopathy (Nervous system disorders) | NA | NA | 0 | 1
Sciatica (Nervous system disorders) | NA | NA | 0 | 1
Seizure (Nervous system disorders) | NA | NA | 2 | 6
Spinal cord haemorrhage (Nervous system disorders) | NA | NA | 0 | 1
Status epilepticus (Nervous system disorders) | NA | NA | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | NA | NA | 1 | 2
Subdural hygroma (Nervous system disorders) | NA | NA | 1 | 0
Syncope (Nervous system disorders) | NA | NA | 36 | 30
Transient ischaemic attack (Nervous system disorders) | NA | NA | 9 | 10
Vertebrobasilar insufficiency (Nervous system disorders) | NA | NA | 0 | 1
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | NA | NA | 1 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | NA | NA | 1 | 0
Device breakage (Product Issues) | NA | NA | 0 | 2
Device defective (Product Issues) | NA | NA | 0 | 1
Device dislocation (Product Issues) | NA | NA | 1 | 0
Device failure (Product Issues) | NA | NA | 0 | 1
Device fastener issue (Product Issues) | NA | NA | 0 | 1
Device malfunction (Product Issues) | NA | NA | 0 | 1
Device occlusion (Product Issues) | NA | NA | 1 | 0
Lead dislodgement (Product Issues) | NA | NA | 1 | 1
Anxiety (Psychiatric disorders) | NA | NA | 2 | 5
Completed suicide (Psychiatric disorders) | NA | NA | 0 | 1
Confusional state (Psychiatric disorders) | NA | NA | 1 | 2
Delirium (Psychiatric disorders) | NA | NA | 0 | 1
Delusion (Psychiatric disorders) | NA | NA | 1 | 0
Depression (Psychiatric disorders) | NA | NA | 1 | 2
Depression suicidal (Psychiatric disorders) | NA | NA | 0 | 1
Disorientation (Psychiatric disorders) | NA | NA | 1 | 2
Hallucination (Psychiatric disorders) | NA | NA | 0 | 1
Intentional self-injury (Psychiatric disorders) | NA | NA | 1 | 1
Major depression (Psychiatric disorders) | NA | NA | 0 | 1
Mental status changes (Psychiatric disorders) | NA | NA | 2 | 2
Personality change due to a general medical condition (Psychiatric disorders) | NA | NA | 1 | 0
Psychiatric decompensation (Psychiatric disorders) | NA | NA | 1 | 0
Restlessness (Psychiatric disorders) | NA | NA | 1 | 0
Suicidal ideation (Psychiatric disorders) | NA | NA | 2 | 1
Acute kidney injury (Renal and urinary disorders) | NA | NA | 37 | 30
Anuria (Renal and urinary disorders) | NA | NA | 1 | 0
Azotaemia (Renal and urinary disorders) | NA | NA | 0 | 1
Bladder tamponade (Renal and urinary disorders) | NA | NA | 1 | 0
Calculus bladder (Renal and urinary disorders) | NA | NA | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | NA | NA | 5 | 1
Dysuria (Renal and urinary disorders) | NA | NA | 1 | 0
End stage renal disease (Renal and urinary disorders) | NA | NA | 0 | 1
Haematuria (Renal and urinary disorders) | NA | NA | 9 | 7
Haemorrhage urinary tract (Renal and urinary disorders) | NA | NA | 0 | 1
Hydronephrosis (Renal and urinary disorders) | NA | NA | 3 | 2
Nephrolithiasis (Renal and urinary disorders) | NA | NA | 1 | 3
Nephrotic syndrome (Renal and urinary disorders) | NA | NA | 0 | 1
Renal colic (Renal and urinary disorders) | NA | NA | 1 | 0
Renal failure (Renal and urinary disorders) | NA | NA | 10 | 8
Renal haematoma (Renal and urinary disorders) | NA | NA | 1 | 1
Renal impairment (Renal and urinary disorders) | NA | NA | 14 | 6
Ureteric obstruction (Renal and urinary disorders) | NA | NA | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | NA | NA | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | NA | NA | 2 | 1
Urethral obstruction (Renal and urinary disorders) | NA | NA | 0 | 1
Urethral stenosis (Renal and urinary disorders) | NA | NA | 2 | 0
Urinary bladder polyp (Renal and urinary disorders) | NA | NA | 1 | 0
Urinary retention (Renal and urinary disorders) | NA | NA | 6 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | NA | NA | 4 | 1
Breast necrosis (Reproductive system and breast disorders) | NA | NA | 0 | 1
Breast pain (Reproductive system and breast disorders) | NA | NA | 1 | 0
Cervical polyp (Reproductive system and breast disorders) | NA | NA | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | NA | NA | 1 | 0
Hysterocele (Reproductive system and breast disorders) | NA | NA | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | NA | NA | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | NA | NA | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | NA | NA | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | NA | NA | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | NA | NA | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | NA | NA | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | NA | NA | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | NA | NA | 19 | 13
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | NA | NA | 7 | 5
Asphyxia (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | NA | NA | 2 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | NA | NA | 14 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | NA | NA | 34 | 28
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | NA | NA | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | NA | NA | 6 | 2
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | NA | NA | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | NA | NA | 1 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | NA | NA | 1 | 4
Haemothorax (Respiratory, thoracic and mediastinal disorders) | NA | NA | 1 | 2
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | NA | NA | 4 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | NA | NA | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 | 3
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | NA | NA | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | NA | NA | 2 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | NA | NA | 1 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | NA | NA | 4 | 6
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | NA | NA | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | NA | NA | 2 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 | 2
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | NA | NA | 8 | 5
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | NA | NA | 2 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | NA | NA | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | NA | NA | 12 | 13
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | NA | NA | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | NA | NA | 11 | 11
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | NA | NA | 1 | 0
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | NA | NA | 4 | 5
Decubitus ulcer (Skin and subcutaneous tissue disorders) | NA | NA | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | NA | NA | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | NA | NA | 6 | 3
Diabetic wound (Skin and subcutaneous tissue disorders) | NA | NA | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | NA | NA | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | NA | NA | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | NA | NA | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | NA | NA | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | NA | NA | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | NA | NA | 3 | 0
Symmetrical drug-related intertriginous and flexural exanthema (Skin and subcutaneous tissue disorders) | NA | NA | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | NA | NA | 1 | 0
Alcoholic (Social circumstances) | NA | NA | 1 | 0
Immobile (Social circumstances) | NA | NA | 0 | 1
Imprisonment (Social circumstances) | NA | NA | 0 | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | NA | NA | 0 | 1
Transcatheter aortic valve implantation (Surgical and medical procedures) | NA | NA | 0 | 1
Aneurysm ruptured (Vascular disorders) | 0 | 0 | 0 | 1
Angiodysplasia (Vascular disorders) | 0 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 0 | 2 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 3
Aortic occlusion (Vascular disorders) | 0 | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Arterial haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 0 | 2 | 2
Arterial stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Arterial thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 1
Brachiocephalic arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 3
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Distributive shock (Vascular disorders) | 0 | 0 | 1 | 0
Embolism arterial (Vascular disorders) | 0 | 0 | 1 | 0
Extremity necrosis (Vascular disorders) | 0 | 0 | 4 | 1
Femoral artery aneurysm (Vascular disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 7
Hypertension (Vascular disorders) | 0 | 0 | 6 | 9
Hypertensive crisis (Vascular disorders) | 0 | 0 | 4 | 3
Hypertensive emergency (Vascular disorders) | 0 | 0 | 1 | 1
Hypertensive urgency (Vascular disorders) | 0 | 0 | 2 | 2
Hypotension (Vascular disorders) | 0 | 0 | 37 | 15
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 2 | 1
Iliac artery occlusion (Vascular disorders) | 0 | 0 | 1 | 2
Iliac artery stenosis (Vascular disorders) | 0 | 0 | 1 | 0
Intermittent claudication (Vascular disorders) | 0 | 0 | 1 | 3
Ischaemic limb pain (Vascular disorders) | 0 | 0 | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Obstructive shock (Vascular disorders) | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 5 | 3
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 7 | 9
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 0 | 2
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 3 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 3 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 3 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 6 | 9
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 4 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1
Reperfusion injury (Vascular disorders) | 0 | 0 | 1 | 0
Subclavian artery occlusion (Vascular disorders) | 0 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1 | 0
Venous aneurysm (Vascular disorders) | 0 | 0 | 0 | 1
Venous haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 Pre-treatment (N=0) | Ramipril Pre-treatment (N=0) | LCZ696 (N=2820) | Ramipril (N=2816)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 130 | 123
Angina pectoris (Cardiac disorders) | 0 | 0 | 125 | 140
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 85 | 87
Cardiac failure (Cardiac disorders) | 0 | 0 | 128 | 150
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 42 | 57
Constipation (Gastrointestinal disorders) | 0 | 0 | 70 | 99
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 227 | 179
Nausea (Gastrointestinal disorders) | 0 | 0 | 93 | 101
Asthenia (General disorders) | 0 | 0 | 67 | 58
Fatigue (General disorders) | 0 | 0 | 125 | 136
Non-cardiac chest pain (General disorders) | 0 | 0 | 183 | 156
Oedema peripheral (General disorders) | 0 | 0 | 122 | 125
Nasopharyngitis (Infections and infestations) | 0 | 0 | 107 | 72
Pneumonia (Infections and infestations) | 0 | 0 | 58 | 66
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 54 | 57
Urinary tract infection (Infections and infestations) | 0 | 0 | 97 | 95
Blood creatinine increased (Investigations) | 0 | 0 | 51 | 58
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 256 | 249
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 76 | 56
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 114 | 103
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 72 | 103
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 70 | 80
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 88 | 95
Dizziness (Nervous system disorders) | 0 | 0 | 280 | 241
Headache (Nervous system disorders) | 0 | 0 | 78 | 69
Syncope (Nervous system disorders) | 0 | 0 | 52 | 57
Insomnia (Psychiatric disorders) | 0 | 0 | 53 | 74
Renal failure (Renal and urinary disorders) | 0 | 0 | 58 | 50
Renal impairment (Renal and urinary disorders) | 0 | 0 | 124 | 129
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 239 | 359
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 185 | 251
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 63 | 51
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 60 | 79
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 72 | 59
Hypertension (Vascular disorders) | 0 | 0 | 96 | 143
Hypotension (Vascular disorders) | 0 | 0 | 447 | 288
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 66 | 32

LIMITATIONS AND CAVEATS:
In this study there were 25 patients who did not take study treatment after randomization, and thus were not included in the safety set.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-05-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT02924727/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT02924727/SAP_001.pdf